CLINICAL TRIAL: NCT04541693
Title: Early Stability Assessment of the REDAPT Revision Hip System With Radiostereometric Analysis
Brief Title: REDAPT Revision Hip System With RSA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic Innovation Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018-092
Record Dates: First submitted 2020-08-31; First posted 2020-09-09 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hip revision (Other): Revision to cup and stem, cup only or stem only.
  Interventions: Device: Full revision; Device: Cup revision; Device: Stem revision

INTERVENTIONS:
Device: Full revision — Both cup and stem require revision
Device: Cup revision — Only the cup requires revision
Device: Stem revision — Only the stem requires revision

SUMMARY:
The principal objectives of the study are to evaluate early and mid-term fixation of the REDAPT revision hip stem and acetabular cup as measured by stem subsidence and proximal cup migration at 2 and 5 years post-surgery through model-based RSA. Secondary objectives include; evaluate the progression of migration between 1 and 2 years and between 2 and 5 years, assess pre- to post-surgery patient improvement in function and health status, evaluate femoral and acetabular radiolucency at 2 and 5 years, and assess patterns of stem migrate on for different revision scenarios (preservation of the trochanters and extended trochanteric osteotomy).

DETAILED DESCRIPTION:
This is a prospective, single arm, consecutive series study of patients undergoing revision hip arthroplasty. Patients will be grouped based on the revision implants they receive during surgery. Patients who receive a full hip revision (stem and cup), will be counted in both study groups. The two study groups are:

1. femoral stem revision (n=30 hips)
2. acetabular cup revision (n=22 hips)

ELIGIBILITY:
Inclusion Criteria:

* Patients needing revision hip arthroplasty in which either the femoral stem or the acetabular cup, or both components, will be revised
* Ability to use study device (not requiring specialized implants)
* Patients between the ages of 18+ older
* Patients willing and able to comply with follow-up requirements and self-evaluations
* Ability to give informed consent

Exclusion Criteria:

* Acute infection requiring washout, debridement, and liner exchange
* Unresolved infection
* Undergoing stage 1 of a 2-stage revision for infection
* Known metal allergy to device components
* Active participation in another clinical study (within the past 30 days)
* Known risk for loss to follow-up (significant geographical distance from treatment centre)
* BMI>40 (severe obesity)
* Unable to provide informed consent (cognitive impairment)
* Patients requiring a bearing couple different than metal on polyethylene
* Patients requiring extreme distal press-fit revision stems (greater than 240 mm in length)
* Patients with severe defects, dysplasia, or tumor
* Inflammatory joint disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in RSA Migrations from baseline(2-week) to 6-month, 1-year and 2-year | Post-op: 2-week, 6-month, 1-year, 2-year
  Stability over a period of two year measured by migration with Röntgen Stereometric Analysis
Changes in Oxford-12 Hip Score from baseline(pre-op) to 6-month, 1-year and 2-year | Pre-op, Post-op (6 months, 1 year, and 2 years)
  The Oxford Hip Score (OHS) is a patient self-administered 12-item questionnaire with each question having a Likaert-like response option. Each item is scored from 0 to 4, and the items are summated, with lower total scores indicating poorer performance. The OHS measures pain and general activities of daily living.
Changes in EQ-5D-5L from baseline(pre-op) to 6-month, 1-year and 2-year | Pre-op, Post-op (6 months, 1 year, and 2 years)
  The EuroQol 5D 5L questionnaire is a standardized instrument for use as a measure of health outcome that is designed for completion by the subject.
Change is Pain VAS from baseline(pre-op) to 6-month, 1-year and 2-year | Pre-op, Post-op (6 months, 1 year, and 2 years)
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in patient reported satisfaction as measured using the visual analogue scale (VAS) from 0 (No pain) - 100 (Worst pain imaginable)
Changes in Patient Satisfaction (Likert scale) from baseline(pre-op) to 6-month, 1-year and 2-year | Pre-op, Post-op (6 months, 1 year, and 2 years)
  Patient satisfaction with their hip surgery will be assessed using a 5-point Likert scale: Very Unsatisfied (1), Unsatisfied (2), Neutral (3), Satisfied (4), and Very Satisfied (5).

SECONDARY OUTCOMES:
Stem subsidence | 1-year, 2-year
  Comparing RSA exams at the specified time points to determine relative movement of the REDAPT hip stem

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Turgeon, MD, Principal Investigator — Concordia Joint Replacement Group
Locations (1):
- Concordia Hospital, Winnipeg, Manitoba, Canada